CLINICAL TRIAL: NCT06439498
Title: Frequency of Orthostatic Hypotension and Affecting Factors in Patients Who Underwent Colonoscopy with Procedural Sedoanalgesia
Brief Title: Frequency of Orthostatic Hypotension in Patients Who Underwent Colonoscopy
Status: Active, not recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Gülencan Yumuşak Ergin, Specialist, Ankara University
Other Study IDs: 109-SBKAEK
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-05

CONDITIONS: Orthostatic Hypotension
Keywords: orthostatic hypotension; colonoscopy
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Patients who will undergo colonoscopy accompanied by sedoanalgesia will be admitted at Aksaray Training and Research Hospital Gastroenterology Clinic between May and July 2024. Orthostatic hypotension will be evaluated after patients meet the discharge criteria in the postoperative recovery unit.

DETAILED DESCRIPTION:
Patients over the age of 18 who apply to the endoscopy unit for colonoscopy will be included. Patients who will be excluded from the study; Patients with cognitive dysfunction for whom consent could not be obtained Patients who cannot walk

Routine ASA (American Society of Anesthesiologist) monitoring will be applied when patients are taken to the procedure room. Patients will be monitored for oxygen saturation with an oxygen saturation probe, non-invasive blood pressure monitoring, and heart rate and rhythm monitoring with an electrocardiogram. Patients will be given oxygen support via nasal cannula or mask. Patients will be given maintenance intravenous fluids. Patients will receive moderate to deep sedation/analgesia. At the end of the procedure, patients will be taken to the postoperative recovery unit and monitored. Patients will be evaluated according to the Aldrete score and a discharge decision will be made. When the decision to discharge the patients is made, they will first be seated and vital signs will be monitored when they are first placed in a sitting position and at the 3rd minute in the sitting position. Then, the patients will be stood up and vital signs will be monitored when they first stand up and at the 3rd minute. It will be noted whether patients develop additional symptoms. Patients who do not have symptoms and are decided to be discharged will be taken to a second waiting room and will be monitored under observation for a while.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who apply to the endoscopy unit for colonoscopy will be included.

Exclusion Criteria:

* Patients with cognitive dysfunction for whom consent could not be obtained Patients who cannot walk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo colonoscopy accompanied by sedoanalgesia will be admitted at Aksaray Training and Research Hospital Gastroenterology Clinic between May and July 2024.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Non invasive blood pressure when sitting position | during first 3 minutes after sitting
  Non invasive blood pressure when sitting position
Non invasive blood pressurewhen standing position | during first 3 minutes after standing
  Non invasive blood pressure when standing position

CONTACTS AND LOCATIONS:
Overall Officials: Gülencan YUMUŞAK ERGİN, Principal Investigator — Ankara University
Locations (1):
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)